CLINICAL TRIAL: NCT02978820
Title: Core Stabilization Exercise Versus Scientific Exercises Approach to Scoliosis in the Treatment of Adolescent Idiopathic Scoliosis: A Randomized Single Blind Trial
Brief Title: The Comparison of Core Stabilization Exercise With Scientific Exercise Approach to Scoliosis in Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Gözde Gür, Research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO 16/82
Record Dates: First submitted 2016-11-20; First posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Scoliosis; Adolescent Idiopathic Scoliosis
Keywords: scientific exercise approach to scoliosis; core stabilization training; bracing; adolescent idiopathic scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEAS exercise group (Experimental): This group received SEAS exercises in addition to brace wearing for four months
  Interventions: Other: SEAS exercise
- CS exercise group (Experimental): This group received core stabilization exercise training (CS) in addition to brace wearing for four months
  Interventions: Other: CS exercise

INTERVENTIONS:
Other: SEAS exercise — Patient were referred by medical doctor with a prescription of brace and exercise training for their moderate scoliotic curves. Patients were randomly divided into two groups. The SEAS group received SEAS exercises one times in a week for four months. In addition patients in SEAS groups were wearing spinal brace for their scoliosis in this period
  Arms: SEAS exercise group
Other: CS exercise — Patient were referred by medical doctor with a prescription of brace and exercise training for their moderate scoliotic curves. Patients were randomly divided into two groups. The CS group received core stabilization exercise training one times in a week for four months. In addition patients in SEAS groups were wearing spinal brace for their scoliosis in this period
  Arms: CS exercise group

SUMMARY:
Scoliosis specific exercises have been shown to improve curve progression but there have been few studies that compare the different exercise approaches in adolescent idiopathic scoliosis (AIS). The objective of this study was to compare the effects of Core stabilization (CS) exercises with Scientific Exercises Approach to Scoliosis (SEAS exercises) in addition to brace wearing in patients with AIS. It is important to compare different exercise methods on different aspects of scoliotic deformity, such as curve progression, angle of trunk rotation, body symmetry, cosmetic trunk deformity, satisfaction with treatment and quality of life.

DETAILED DESCRIPTION:
The aim of this study was to investigate whether adolescent with idiopathic scoliosis receiving scoliosis specific exercise approach, such as SEAS exercises, in accordance with the bracing approach for moderate curves would have greater improvement in curve progression, trunk deformity, body symmetry and quality of life than adolescent receiving exercise therapy based on the general core stabilization approach with similar intensity. Thirty female patients with AIS aged 12 to16 years, who have moderate curves (20 to 45 degree) randomly divided into two groups. One group received CS exercise, while other received SEAS exercise for forty-min once weekly for four months. Both groups underwent full-time bracing (23 hours per day) intervention. Outcome was based on Cobb angle, angle of trunk rotation, body symmetry (Posterior Trunk Symmetry Index), cosmetic trunk deformity (Walter Reed Visual Assessment Scale) and quality of life (Scoliosis Research Society - 22 Questionnaire) measured at baseline and after intervention period. Results were analyzed using the paired sample t-test to compare repeated measurements and independent sample t-test to compare the groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in the current study were consecutive adolescents with idiopathic scoliosis seen in our department who were referred to receive both brace and exercise treatment conservatively. Additional inclusion criteria included the following: female gender; at least age 12 years; primary curve magnitude between 20 and 45 degrees of Cobb angle; double curve (right thoracic-left lumbar) or single thoracolumbar curve having an apex in the main thoracic region; Risser 2-3 and no previous treatment.

Exclusion Criteria:

* Exclusion criteria for both groups were as follows: evidence of congenital curve; neuromuscular, rheumatologic, renal, cardiovascular, pulmonary or vestibular diseases or surgical correction history.

Ages: 12 Years to 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Cobb angle | Change from baseline Cobb angle at 4 months
  Cobb angle is considered a gold standard to determine the magnitude of spinal curve on frontal plan radiograph

SECONDARY OUTCOMES:
Chance in Posterior trunk symmetry index | Change from baseline trunk symmetry at 4 months
  Posterior trunk symmetry index includes the sensitive assessment of the frontal plane asymmetry of trunk deformity as a two-dimensional surface topographic method in scoliosis. The index based on assessing trunk asymmetry with regard to C7 plumb line, shoulder and hip asymmetry based on back surface photograph of patient.
Change in Walter reed visual assessment scale | Change from baseline cosmetic trunk deformity at 4 months
  Walter reed visual assessment scale assesses patient's cosmetic trunk deformity with set of figures representing seven visible aspects of spinal deformity: Item 1, spinal deformity; item 2, rib prominence; item 3, lumbar prominence; item 4, thoracic deformity; item 5, trunk imbalance; item 6, shoulder asymmetry; and item 7, scapular asymmetry
Change in Scoliosis Research Society 22 Questionnaire | Change from baseline quality of life at 4 months
  Scoliosis Research Society 22 Questionnaire is widely used to evaluate the efficacy of several treatment regimens for idiopathic scoliosis from the patient's perception of his or her condition. The questionnaire consists of 22 items exploring 5 domains related to psychophysical wellbeing: function/activity level, pain, mental health, self-image and treatment satisfaction.
Change in Angle of trunk rotation | Change from baseline angle of trunk rotation at 4 months
  Angle of Trunk rotation is assessed with scoliometer in forward bending test

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Negrini S, Aulisa AG, Aulisa L, Circo AB, de Mauroy JC, Durmala J, Grivas TB, Knott P, Kotwicki T, Maruyama T, Minozzi S, O'Brien JP, Papadopoulos D, Rigo M, Rivard CH, Romano M, Wynne JH, Villagrasa M, Weiss HR, Zaina F. 2011 SOSORT guidelines: Orthopaedic and Rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis. 2012 Jan 20;7(1):3. doi: 10.1186/1748-7161-7-3. PMID 22264320
- [Background] Negrini S, Grivas TB, Kotwicki T, Maruyama T, Rigo M, Weiss HR; Members of the Scientific society On Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT). Why do we treat adolescent idiopathic scoliosis? What we want to obtain and to avoid for our patients. SOSORT 2005 Consensus paper. Scoliosis. 2006 Apr 10;1:4. doi: 10.1186/1748-7161-1-4. PMID 16759352
- [Background] Weinstein SL. Adolescent idiopathic scoliosis: prevalence and natural history. Instr Course Lect. 1989;38:115-28. PMID 2649564
- [Background] Smania N, Picelli A, Romano M, Negrini S. Neurophysiological basis of rehabilitation of adolescent idiopathic scoliosis. Disabil Rehabil. 2008;30(10):763-71. doi: 10.1080/17483100801921311. PMID 18432434
- [Background] Fusco C, Zaina F, Atanasio S, Romano M, Negrini A, Negrini S. Physical exercises in the treatment of adolescent idiopathic scoliosis: an updated systematic review. Physiother Theory Pract. 2011 Jan;27(1):80-114. doi: 10.3109/09593985.2010.533342. PMID 21198407
- [Background] Romano M, Negrini A, Parzini S, Tavernaro M, Zaina F, Donzelli S, Negrini S. SEAS (Scientific Exercises Approach to Scoliosis): a modern and effective evidence based approach to physiotherapic specific scoliosis exercises. Scoliosis. 2015 Feb 5;10:3. doi: 10.1186/s13013-014-0027-2. eCollection 2015. PMID 25729406
- [Background] Gur G, Ayhan C, Yakut Y. The effectiveness of core stabilization exercise in adolescent idiopathic scoliosis: A randomized controlled trial. Prosthet Orthot Int. 2017 Jun;41(3):303-310. doi: 10.1177/0309364616664151. Epub 2016 Sep 13. PMID 27625122